CLINICAL TRIAL: NCT05803512
Title: Predicting Female Pelvic Tilt and Lumbar Angle Using Machine Learning in Case of Urinary Incontinence and Sexual Dysfunction
Status: Completed | Type: Observational
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Other Study IDs: 1\2023
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: The Purpose of This Study is to Predicting Female Pelvic Tilt and Lumbar Angle Using Machine Learning in Case of Urinary Incontinence and Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: urinary incontinence females with sexual dysfunction
- control group: Normal females

SUMMARY:
The purpose of this study is to Predicting female pelvic tilt and lumbar angle using machine learning in case of urinary incontinence and sexual dysfunction

DETAILED DESCRIPTION:
92 patients were distributed randomly into two groups. The first group will be measured pelvic tilt, lumbar angle by spinal mouse and force of contraction of pelvic floor muscles by ultrasound imaging, UDI-6 and FSFI questionnaires for urinary incontinence female The second group will be measured pelvic tilt, lumbar angle by spinal mouse device and force of contraction of pelvic floor muscles by ultrasound imaging, UDI-6 and FSFI questionnaires for normal females.

Patients will be examined by radiologist with medical ultrasound imaging and by me with spinal mouse device.

ELIGIBILITY:
Inclusion Criteria:

* - Their ages varied from 30to 40years, their body mass index (BMI) was 25-30 kg/m2 and a number of parities ≤ three normal vaginal deliveries, at least two years and Subjects hadn't received drugs, patients with mild and moderate urinary incontinence with sexual dysfunction

Exclusion Criteria:

- 1. History of spinal surgery or spinal fracture. 2. Volunteers with a history of a recto-vaginal or vesico-vaginal fistula, undiagnosed uterine bleeding urinary tract infection, diabetes, intrauterine device, chest and/or cardiac disease and using any drugs for urinary incontinence 3. Serious diseases, such as heart disease, kidney, liver diseases, gastric ulcer or duodenal ulcer.

4. A history of bronchial asthma or any chest disease. 5. Uncontrolled diabetes or hypertension. 6. Patients with peacemaker or any metal implant on the treated area. 7. Cancer or patient with past history of tumor excision.

Ages: 30 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Their ages varied from 30to 40years, their body mass index (BMI) was 25-30 kg/m2 and a number of parities ≤ three normal vaginal deliveries
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Pelvic tilt, lumbar angle | 2 months
  by spinal mouse device evaluation was carried out with the individuals standing erect and in the maximum trunk flexion and extension postures. The sagittal curvatures of the thoracic spine (T1-2 to T11-12) and lumbar spine (T12-L1 to the sacrum) were measured, as well as the position of the sacrum and hips (difference between the sacral angle and the vertical position).

SECONDARY OUTCOMES:
Force of contraction of pelvic floor muscles | 2 months
  muscles by ultrasound imaging, convex transducer was used at a frequency of 5 MHz for evaluating. Voluntary PFM contractions' force (strength) of all patients

CONTACTS AND LOCATIONS:
Overall Officials: tarek Abd Elhafez, Principal Investigator — Deraya University
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No